CLINICAL TRIAL: NCT05525754
Title: Effectiveness of Computed Tomography-Guided Nasotracheal Intubation Procedure on Predicting Tube Advancement Difficulty and Preventing Epistaxis: A Prospective Case-control Study
Brief Title: Computed Tomography-Guided Nasotracheal Intubation Procedure
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, seher orbay yasli, Assistant Professor, TC Erciyes University
Other Study IDs: 2018 /No:377
Record Dates: First submitted 2022-08-29; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Computed Tomography-guided Nasotracheal Intubation; The Space Where the Tube Will be Passed in the Internal Nasal Valve Region
Keywords: Computed Tomography; epistaxis; Maxillofacial Orthognathic Surgery; Intubation
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: computed tomography-guided nasotracheal intubation — Before intubation, the lower part of the nasal valve region, aka the narrowest area of the nasal passage, was measured by calculating the distance between the anterior border of the inferior concha and the septal cartilage

SUMMARY:
Background: Nasotracheal intubation can lead to severe complications like epistaxis with excessive bleeding. The advancement difficulty of the tube faced during nasal intubation is one of the fundamental causes of this condition. The present study aimed to evaluate the effectiveness of Computed tomography-guided nasotracheal intubation in predicting tube advancement difficulty and preventing epistaxis.

Material and Methods: 60 maxillofacial surgery patients were included in the study. The space where the tube will be passed in the internal nasal valve region was measured horizontally (distance between inferior concha and septum) and vertically (distance between inferior concha and hard palate) by Computed Tomography. The patients were divided into two groups, 'easy' (n=28) or 'difficult' (n=32), according to the effort required to advance the tube through the nasal passage.

ROC analysis was performed, and cut-off values were determined to reveal the distance values at which difficulty may be experienced while advancing the tube. The cut-off values were 1.09 cm and 0.39 cm for the vertically and horizontally distances, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 who underwent bimaxillary orthognathic surgery
* defined as ASA (American Society of Anesthesiology) I or II

Exclusion Criteria:

* The lack of preoperative CT scans
* airways evaluated and considered difficult by the anesthesiologist
* airways assessed and considered not appropriate for right angle endotracheal (RAE) tube with7.0 mm internal diameter
* history of sinusitis or head trauma
* anticoagulant therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sixty health volunteers who went orthognathic surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Investigation of the relationship between internal nasal valve measurements and nasal advancement of the intubation tube | during intubation procedure
  The measurements were carried out from the coronal sections at 0.25 intervals. Before intubation, the lower part of the nasal valve region, aka the narrowest area of the nasal passage, was measured by calculating the distance between the anterior border of the inferior concha and the septal cartilage. Additionally, using the same section of the CT image, the distance between the inferior concha and the hard palate was measured

CONTACTS AND LOCATIONS:
Overall Officials: SEHER Orbay Yaşlı, Principal Investigator — Erciyes University Faculty of Dentistry
Locations (1):
- SEHER Orbay Yaşlı, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yasli SO, Canpolat DG, Baydan E, Demirbas AE. Effectiveness Of Computed Tomography-Guided Nasotracheal Intubation Procedure On Predicting Tube Advancement Difficulty And Preventing Epistaxis: A Prospective Case-Control Study. J Pak Med Assoc. 2023 Oct;73(10):1981-1986. doi: 10.47391/JPMA.8034. PMID 37876056